CLINICAL TRIAL: NCT04003038
Title: A Randomized, Prospective Evaluation of Negative Pressure Wound Therapy on Abdominal Donor Site in Free Flap Breast Reconstruction in Obese Patients
Brief Title: Negative Pressure Wound Therapy in Healing Abdominal Incision in Obese Patients Undergoing Breast Reconstruction Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018-0004; NCI-2019-02777 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0004 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2019-06-27; First posted 2019-07-01 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Body Mass Index Greater Than or Equal to 30; Malignant Breast Neoplasm; Mammoplasty Patient; Obesity
MeSH Terms: conditions — Breast Neoplasms; Obesity | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (wound care with a standard dressing) (Active Comparator): Patients receive wound care with a standard dressing (bandage) after surgery for 7 days.
  Interventions: Procedure: Wound Care Management
- Group II (NPWT) (Experimental): Patients receive NPWT after surgery for 7 days.
  Interventions: Procedure: Negative Pressure Wound Therapy

INTERVENTIONS:
Procedure: Negative Pressure Wound Therapy — Receive wound care with NPWT
  Other Names: NPWT; Vacuum-Assisted Wound Closure
  Arms: Group II (NPWT)
Procedure: Wound Care Management — Receive wound care with a standard dressing (bandage)
  Other Names: Wound Care; Wound Care Treatment; Wound Management; Wound Treatment
  Arms: Group I (wound care with a standard dressing)

SUMMARY:
This trial studies the safety and how well negative pressure wound therapy works in healing the abdominal incision in obese patients undergoing free flap breast reconstruction surgery. Using negative pressure wound therapy (NPWT) instead of standard dressing (bandages) may improve wound healing at the surgical site in the abdomen where tissue was collected for breast reconstruction surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the impact of negative pressure wound therapy on wound healing as measured by wound dehiscence rate.

II. Long-term follow-up on wound healing complications.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive wound care with a standard dressing (bandage) after surgery for 7 days.

GROUP II: Patients receive negative pressure wound therapy (NPWT) after surgery for 7 days.

After completion of study, patients are followed up at 2 weeks, and at 1 and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a free abdominal flap, including a superficial inferior epigastric artery (SIEA), deep inferior epigastric artery perforator (DIEP), or muscle-sparing transverse rectus abdominus myocutaneous (MS-TRAM) flap for breast reconstruction.
* Patients are willing and able to give consent.
* Body mass index (BMI) greater than or equal to 30.0.

Exclusion Criteria:

* Patients who are unable to provide consent.
* Patients who are suspected or known to be pregnant.
* Known allergy to topical adhesives.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-05-02 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Rate of wound dehiscence | Up to 3 months
  Will measure and compare the wound healing outcomes of patients. All adverse events will be identified, graded for severity and assigned causality, reported to the required entities, and compiled for periodic review. After assigning causality, the principal investigator will decide the course of action for the study participant.
Wound healing complications | Up to 3 months
  Will measure and compare the wound healing outcomes of patients. All adverse events will be identified, graded for severity and assigned causality, reported to the required entities, and compiled for periodic review. After assigning causality, the principal investigator will decide the course of action for the study participant.

CONTACTS AND LOCATIONS:
Overall Officials: Edward H Chang, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org